CLINICAL TRIAL: NCT00674024
Title: A Phase I and Pharmacokinetic Single Agent Study of Pazopanib in Adults With Advanced Malignancies and Varying Degrees of Liver Dysfunction
Brief Title: Pazopanib to Treat Adults With Advanced Cancers and Varying Degrees of Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090003; 09-C-0003; NCT01445496 (obsolete NCT alias)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2013-01-22

CONDITIONS: Neoplasms; Lymphoma
Keywords: Pazopanib; Tyrosine Kinase Inhibitor; Advanced Cancer; Pharmacokinetics; Cancer; Solid Tumor; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — pazopanib

INTERVENTIONS:
Drug: Pazopanib
Drug: Pazopanib (GW786034)(GW786034)

SUMMARY:
Background:

* Pazopanib is an experimental drug that was designed to enter cancer cells and block the activity of proteins that are important for cancer cell growth and survival.
* This is the first study in which pazopanib is given to patients with different degrees of liver function. The safe dose for patients with normal liver function is already known.

Objectives:

* To determine the safety and side effects of pazopanib given at different dose levels to patients with cancer who have different degrees of liver function.
* To find out how much pazopanib is in the blood at specific times.
* To determine if pazopanib is effective in treating advanced cancer in patients with different degrees of liver function.

Eligibility:

- Patients 18 years of age and older with an advanced solid tumor or lymphoma that cannot be treated successfully with standard therapies and who have normal or abnormal liver function.

Design:

* Treatment:
* Patients are divided into 4 groups, based on their liver function. The first three patients in each group receive a low dose of pazopanib. The next three in each group receive a higher dose of pazopanib if no serious side effects were reported in the previous three. The dose is increased in succeeding groups of three patients until the maximum study dose is reached.
* Patients take pazopanib once a day by mouth in 21-day treatment cycles. Treatment continues until the cancer worsens, the patient develops severe side effects, the patient no longer wants to continue the study, or the doctor removes the patient from the study for other reasons.
* Monitoring:
* Blood pressure: Patients monitor and record their blood pressure twice a day after starting treatment.
* Blood tests: Patients have weekly routine blood tests. In addition, at week 3 of the first cycle and again after the highest safe dose has been determined, several blood samples are collected at frequent intervals to determine how the body handles the drug.
* Imaging studies: X-rays or scans or both are done to measure the extent of disease every 3 cycles.
* Physical examinations are done at periodic intervals.

DETAILED DESCRIPTION:
Background:

* Pazopanib is a potent, multi-targeted receptor tyrosine kinase inhibitor of VEGFR-1, VEGFR-2, VEGFR-3, PDGFR-alpha, PDGFR-beta, and c-kit with the potential to inhibit angiogenesis, lymphangiogenesis, and tumor growth that may have an advantage over agents with a narrower kinase specificity profile.
* Pazopanib has shown activity in renal cell cancer with tumor shrinkage and stable disease; Phase I, II, and III trials as single therapy and in combination with lapatinib are ongoing or planned in patients with various solid tumors.
* Pazopanib appears to be well tolerated at doses from 50 mg three times weekly to 2000 mg daily; the most common adverse events are hypertension, diarrhea, nausea, fatigue, and hair depigmentation.

Objectives:

* To establish the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of pazopanib in groups of patients with varying degrees of hepatic dysfunction (mild, moderate, and severe) in order to provide appropriate dosing recommendations for pazopanib in such patients.
* To characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profiles of pazopanib and metabolites (GSK1071306, GSK1268992, GSK1268997, and GW700201) in patients with varying degrees of hepatic dysfunction.
* To document the non-DLTs associated with administration of pazopanib in patients with hepatic dysfunction.
* To explore correlations of the Child-Pugh classification of hepatic dysfunction with the observed toxicities, plasma PK, and PD of pazopanib administration.
* To document any antitumor activity associated with pazopanib treatment of patients enrolled on this study.

Eligibility:

* Adult patients must have histologically or cytologically confirmed solid tumor or lymphoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients must have adequate renal and bone marrow function.

Study Design:

* Patients will be stratified into four cohorts according to their hepatic function.
* Pazopanib will be administered orally once daily on days 1-21 of a 21-day cycle.
* Blood samples for PK will be collected from all patients.
* A minimum of 2 and a maximum of 12 patients will be accrued in each liver dysfunction group at each dose, with 12 patients entered at the recommended dose level in each group. At least 12 patients will be accrued in the normal liver function group. The estimated maximum accrual is 132 patients, including all centers.

ELIGIBILITY:
* INCLUSION CRITERIA:

For patients at the NCI, histological or cytological confirmation of solid tumor or lymphoma diagnosis will be performed at the NCI Laboratory of Pathology.

EXCLUSION CRITERIA:

Patients who have had prior treatment with pazopanib will not be eligible for this study.

Patients with abnormal liver function except grade 4 AST, grade 4 ALT, and grade 4 bilirubin will be eligible and will be grouped according to the criteria in Section 5.1. For assessing hepatic dysfunction, greater than 35 percent of the total bilirubin must be direct bilirubin.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10-07; Primary Completion 2013-01-22 (Actual); Study Completion 2013-01-22 (Actual)

PRIMARY OUTCOMES:
To establish the MTD and DLT of pazopanib in groups of patients with varying degrees of hepatic dysfunction (mild, moderate, and severe) to provide appropriate dosing recommendations for panzopanib in such patients.

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profiles of pazopanib and metabolites (GSK1071306, GSK1268992, GSK1268997, and GW700201) in patients with varying degrees of hepatic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Conn HO. A peek at the Child-Turcotte classification. Hepatology. 1981 Nov-Dec;1(6):673-6. doi: 10.1002/hep.1840010617. No abstract available. PMID 7308998
- [Background] Conn HO, Resnick RH, Grace ND, Atterbury CE, Horst D, Groszmann RJ, Gazmuri P, Gusberg RJ, Thayer B, Berk D, Wright SC, Vollman R, Tilson DM, McDermott WV, Cohen JA, Kerstein M, Toole AL, Maselli JP, Razvi S, Ishihara A, Stern H, Trey C, O'Hara ET, Widrich W, Aisenberg H, Stansel HC, Zinny M. Distal splenorenal shunt vs. portal-systemic shunt: current status of a controlled trial. Hepatology. 1981 Mar-Apr;1(2):151-60. doi: 10.1002/hep.1840010211. PMID 7026401